CLINICAL TRIAL: NCT07060131
Title: Observe the Effects of Far Infrared Eye Masks on Acupoints Around the Eyes in Patients With Dry Eye Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC1-054
Record Dates: First submitted 2025-03-11; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease (DED)
Keywords: Far Infrared Eye Masks; Dry Eye Disease; Acupoints Around the Eyes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observe the Effects of Far Infrared Eye Masks on Acupoints Around the Eyes in Patients with DED (Experimental)
  Interventions: Device: Far Infrared Eye Masks

INTERVENTIONS:
Device: Far Infrared Eye Masks — Using far-infrared eye masks on the acupoints around the eyes, including Jingming, Taiyang, Sibai, Tongziliao, and Si Zhu Kong to assess whether there is an improvement in the symptomatic indicators of dry eye disease.

SUMMARY:
Dry eye disease (DED) is a multifactorial ocular surface condition characterized by instability of the tear film. DED is common in ophthalmic and optometric clinical practice, and meibomian gland dysfunction (MGD) has been identified as a major cause of evaporative DED. The use of heated eye mask is a common recommendation in the treatment of MGD, aiming to adequately heat the meibum to increase its liquefaction and flow. Several products are available for this purpose (e.g., Bruder Moist Heat Eye Compress [Bruder Healthcare Company], EyeGiene® [Eyedetec Medical], Blepha EyeBag® [formerly MGDRx EyeBag, Théa Pharmaceuticals Ltd], Blephasteam® [Théa Pharmaceuticals Ltd]).

This study employs far-infrared eye masks on the acupoints around the eyes, including Jingming, Taiyang, Sibai, Tongziliao, and Si Zhu Kong to assess whether there is an improvement in the symptomatic indicators of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

*Clinical diagnosis of Dry Eye Disease by Ocular Surface Disease Index (OSDI) ≥ 13 and NIBUT <10 seconds.

Exclusion Criteria:

* Eye inflammation
* Eyelid malposition, such as entropion, ectropion, and upper eyelid ptosis
* Recent eye surgery (within 3 months)
* Risks of retinal detachment such as high myopia, lattice degeneration, and retinal holes
* Use anti-inflammatory eye drops (topical steroids or cyclosporine) within 1 month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Two-tailed Paired T-test of Persons with Dry Eye Diseases with Far Infrared Mask Treatment Assessed by _OSDI | 2 years
  OSDI is collected in scores All the data mentioned above will be collected before and after treatment one month later. They will be compared with two-tailed paired t-test separately. P < 0.05 was considered statistically significant.
Two-tailed Paired T-test of Eyes with Dry Eye Diseases with Far Infrared Mask Treatment Assessed by _NIBUT(non-invasive break-up time) | 2 years
  NIBUT(non-invasive break-up time) recorded in sec will be collected before and after treatment 30 mins and one month later. They will be compared with two-tailed paired t-test separately. P < 0.05 was considered statistically significant.
Two-tailed Paired T-test of Eyes with Dry Eye Diseases with Far Infrared Mask Treatment Assessed by _Meibomian Gland Loss | 2 years
  Meibomian Gland Loss in percentage will be collected before and after treatment 30 mins and one month later . They will be compared with two-tailed paired t-test separately. P < 0.05 was considered statistically significant.
Two-tailed Paired T-test of Eyes with Dry Eye Diseases with Far Infrared Mask Treatment Assessed by _Schirmer test | 2 years
  Description: Schirmer test in mm. All the data mentioned above will be collected before and after treatment 30 mins and one month later. They will be compared with two-tailed paired t-test separately. P < 0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North Dist, Taiwan

REFERENCES:
- [Background] Valencia-Nieto L, Novo-Diez A, Blanco-Vazquez M, Lopez-Miguel A. Therapeutic Instruments Targeting Meibomian Gland Dysfunction. Ophthalmol Ther. 2020 Dec;9(4):797-807. doi: 10.1007/s40123-020-00304-3. Epub 2020 Sep 24. PMID 32968960
- [Background] Sheppard JD, Nichols KK. Dry Eye Disease Associated with Meibomian Gland Dysfunction: Focus on Tear Film Characteristics and the Therapeutic Landscape. Ophthalmol Ther. 2023 Jun;12(3):1397-1418. doi: 10.1007/s40123-023-00669-1. Epub 2023 Mar 1. PMID 36856980
- See also: Related Info — https://www.researchgate.net/publication/356053855_Chambered_warm_moist_air_eyelid_warming_devices_-_a_review#pf7